CLINICAL TRIAL: NCT00400465
Title: Is the Routine Pressure Dressing After Thyroidectomy Necessary? A Prospective Randomized Controlled Study
Brief Title: Is the Routine Pressure Dressing After Thyroidectomy Necessary?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Patorn Piromchai, Department of Otorhinolaryngology, Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE49-1009; ISRCTN52660978 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Neoplasms; Thyroid Nodules; Graves Disease; Goiter
Keywords: thyroid; thyroidectomy; dressing
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Graves Disease; Goiter; Thyroid Diseases | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Pressure dressing
  Interventions: Procedure: Pressure dressing
- Experimental group (Experimental): Normal dressing
  Interventions: Procedure: Normal dressing

INTERVENTIONS:
Procedure: Normal dressing — Normal dressing
  Arms: Experimental group
Procedure: Pressure dressing — Pressure dressing
  Arms: Control group

SUMMARY:
Thyroidectomy is an operation that is commonly performed. After an operation a pressure dressing by Hypafix is usually used due to the belief that it will help to reduce complications such as post-operative bleeding or haematoma. However, the practice is uncomfortable to patients and makes it hard to detect early haematomas.

We carried out a prospective randomised study to study the role of pressure dressing after thyroid surgery by evaluating the amount of fluids collected in the operative bed by ultrasonography compared with normal dressing.

DETAILED DESCRIPTION:
Thyroidectomy is an operation that is commonly performed. In Department of Otolaryngology, Khonkaen University was performed this operation about 200 cases per years. After an operation a pressure dressing by Hypafix is usually used due to the belief that it will help to reduce complications such as post-operative bleeding or haematoma. However, the practice is uncomfortable to patients and makes it hard to detect early haematomas.

We carried out a prospective randomised study to study the role of pressure dressing after thyroid surgery by evaluating the amount of fluids collected in the operative bed by ultrasonography compared with normal dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent thyroidectomy in Srinagarind hospital, Khonkaen University

Exclusion Criteria:

* Patients with cervical lymph nodes metastases requiring neck dissection
* Patients that tissue pathology shown anaplastic carcinoma
* Patients with clinical or laboratory indicators of coagulation disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
amount of fluids collected in the operative bed by ultrasonography | participants will be followed for the duration of hospital stay, an expected average of 4 days

SECONDARY OUTCOMES:
Days retained drains | participants will be followed for the duration of hospital stay, an expected average of 4 days
days of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 4 days
complication (bruise,bleeding,wound dehiscence) | participants will be followed for the duration of hospital stay, an expected average of 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Patorn Piromchai, MD, Principal Investigator — Khonkaen University
Locations (1):
- Deapartment of Otolaryngology, Srinagarind Hospital, Khonkaen University, Muang, Khonkaen, Thailand

REFERENCES:
- [Background] FALCAO P. [Use of compensated pressure dressing in thyroid surgery]. Rev Paul Med. 1951 Jul;39(1):64-6. No abstract available. Undetermined Language. PMID 14865291
- [Background] FALCAO P. [Use of a compressive-compensed dressing in thyroid surgery]. Rev Bras Otorrinolaringol. 1951 May-Jun;19(3A):88-90. No abstract available. Undetermined Language. PMID 14876034
- [Background] Abbas G, Dubner S, Heller KS. Re-operation for bleeding after thyroidectomy and parathyroidectomy. Head Neck. 2001 Jul;23(7):544-6. doi: 10.1002/hed.1076. PMID 11400242
- [Background] Palestini N, Tulletti V, Cestino L, Durando R, Freddi M, Sisti G, Robecchi A. [Post-thyroidectomy cervical hematoma]. Minerva Chir. 2005 Feb;60(1):37-46. Italian. PMID 15902052
- [Background] Cichon S, Anielski R, Orlicki P, Krzesiwo-Stempak K. [Post-thyroidectomy hemorrhage]. Przegl Lek. 2002;59(7):489-92. Polish. PMID 12516234
- [Background] Agarwal A, Mishra SK. Post-thyroidectomy haemorrhage: an analysis of critical factors in successful management. J Indian Med Assoc. 1997 Jul;95(7):418-9, 433. PMID 9425841
- [Background] Shaha AR, Jaffe BM. Practical management of post-thyroidectomy hematoma. J Surg Oncol. 1994 Dec;57(4):235-8. doi: 10.1002/jso.2930570406. PMID 7990478
- [Derived] Piromchai P, Vatanasapt P, Reechaipichitkul W, Phuttharak W, Thanaviratananich S. Is the routine pressure dressing after thyroidectomy necessary? A prospective randomized controlled study. BMC Ear Nose Throat Disord. 2008 Mar 20;8:1. doi: 10.1186/1472-6815-8-1. PMID 18366712